CLINICAL TRIAL: NCT02502474
Title: Study of the Colonic Carriage of Staphylococcus Aureus in a Prospective Cohort of Patients Undergoing Endoscopic Screening for Digestive Cancer in the University Hospital of Saint-Etienne.
Acronym: ColoStaph
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1408023; 2014-A00755-42 (Other: ANSM)
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: STAPHYLOCOCCAL INFECTIONS
Keywords: staphylococcus aureus; digestive carriage; mucosal colonization
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing a colonoscopy (Experimental): Staphylococcus aureus carriage is measured in nose, throat, colon, rectum and groin
  Interventions: Other: Staphylococcus aureus carriage

INTERVENTIONS:
Other: Staphylococcus aureus carriage — nasal, throat, rectal and groin sampling with swabs. Colonic sampling by colonic biopsy

SUMMARY:
Epidemiological study aiming to describe the carriage (nasal, throat, groin, rectal and colonic) of S. aureus in patients without chronic digestive disease who are going to have a colonoscopy for cancer screening. The carriage will be analyzed globally and the similarity of strains isolated from each site will be analyzed using molecular tools. The aim of this study is to better estimate the digestive reservoir of S. aureus to better prevent endogenous infections due to this bacterium.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated to French social security
* Written consent of the patient
* Patient needing a colonoscopy in the University Hospital of Saint-Etienne, France

Exclusion Criteria:

* Patient who decline to participate to the study
* Patient in the incapacity to give consent
* Patient receiving treatment with anticoagulant or antiaggregant platelets
* Patients with a known haemostatic disorder
* Pregnant woman
* Patients with a chronic disease of the gastrointestinal tract
* Patients receiving long-term corticosteroid
* Patient receiving anti staphylococcal antibiotics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Number of patient with Staphylococcus aureus colonic carriage | Day 1
  Staphylococcus aureus carriage in the colon is measured by biopsy

SECONDARY OUTCOMES:
Number of patient with similar Staphylococcus aureus strains in the nose and in the rectum | Day 1
  Staphylococcus aureus carriage in the rectum and in the nose is measured by swab culture
Number of patient with Staphylococcus aureus carriage in the nose | Day 1
  Staphylococcus aureus carriage in the nose is measured by swab culture.
Number of patient with Staphylococcus aureus carriage in the throat | Day 1
  Staphylococcus aureus carriage in the throat is measured by swab culture.
Number of patient with Staphylococcus aureus carriage in the groin | Day 1
  Staphylococcus aureus carriage in the groin is measured by swab culture.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Berthelot, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No